CLINICAL TRIAL: NCT03168464
Title: Radiation and Immune Checkpoints Blockade in Metastatic NSCLC (BMS # CA209-632)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607017434
Record Dates: First submitted 2017-05-19; First posted 2017-05-30 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Ipilimumab; Nivolumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Eligible patients will receive on Day 1 ipilimumab 3mg/kg concurrently with Radiation therapy (6GY x 5 fractions). On Day 22, patients will receive nivolumab 240mg (every 2 weeks) in addition to ipilimumab (1mg/kg). Patients will be evaluated for response at Day 70 (+/- 7 days) for progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Immunotherapy + Radiation (Experimental): Non-ablative radiotherapy (6GyX5) is directed to one lesion during a first immunotherapy treatment with Ipilimumab 3 mg/kg (± 24hrs from first RT dose). On day 22 the combined treatment of ipilimumab plus nivolumab will start (nivolumab 240mg q 2 weeks, ipilimumab 1mg/kg q 6 weeks), and administered until evidence of progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab (3mg/kg) is given concurrently (+/- 24hrs from first RT dose) with radiation therapy on Day 1 of the study. On day 22 the combined treatment of ipilimumab plus nivolumab will start (nivolumab 240mg q 2 weeks, ipilimumab 1mg/kg q 6 weeks), and administered until evidence of progression.
  Other Names: Yervoy
Drug: Nivolumab — On day 22 the combined treatment of ipilimumab plus nivolumab will start (nivolumab 240mg q 2 weeks, ipilimumab 1mg/kg q 6 weeks), and administered until evidence of progression.
  Other Names: OPDIVO
Radiation: Radiation therapy — Ipilimumab (3mg/kg) is given concurrently (+/- 24hrs from first RT dose) with radiation therapy on Day 1 of the study.

SUMMARY:
NSCLC patients with metastatic disease who have failed at least one prior treatment and have a minimum of two metastatic lesions (at least one measurable), are eligible if they have an ECOG Performance Status of 0-1. Patients will receive on Day 1, ipilimumab (every 6 weeks) concurrently with radiation (6Gy x 5 fractions). Nivolumab (every 2 weeks) will be given in addition to ipilimumab on day 22.

DETAILED DESCRIPTION:
NSCLC patients with metastatic disease who have failed at least one prior treatment and have a minimum of two metastatic lesions (at least one measurable), are eligible if they have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.

Non-ablative radiotherapy (6GyX5) is directed to one lesion during a first immunotherapy treatment with Ipilimumab 3 mg/kg (± 24hrs from first RT dose). On day 22 the combined treatment of ipilimumab plus nivolumab will start (nivolumab 240mg q 2 weeks, ipilimumab 1mg/kg q 6 weeks), and administered until evidence of progression.

Patients are re-imaged at Week 9 (day 70 ± 7) to evaluate for response (defined as an objective response by RECIST of the measurable metastatic sites outside the radiation field). This response will be evaluated assessing clinical and positron emission computed tomography (PET/CT) responses in the non-irradiated measurable metastatic sites using RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document;
* Histologic diagnosis of NSCLC;
* Any Kras or epidermal growth factor receptor (EGFR) status is permitted; Patients with an EGFR sensitizing mutation must have received an EGFR tyrosine kinase inhibitor (either erlotinib, gefitinib or afatinib) and patients with anaplastic lymphoma kinase (ALK) translocation must have received anti-ALK therapy.
* Patients must have at least two distinct measurable metastatic sites, with one of at least 1 cm or larger in its largest diameter. Patients may have additional non-measurable metastatic lesions (e.g., bone metastases);
* Patients must have prior treatment with at least one line of therapy for metastatic NSCLC. Any prior therapy is permitted except prior therapy with ipilimumab, other anti cytotoxic T-lymphocyte-associated protein (CTLA) agents or Checkpoint inhibitors;
* An interval of 2 weeks from last previous therapy is required;
* Patients must have recovered from the toxic effect(s) of the most recent anti-cancer treatment to NCI CTCAE Grade 1 or less (except alopecia).
* Patients must have adequate organ and marrow function as defined by initial laboratory tests:

white blood cell (WBC) ≥ 2000/uL

* absolute neutrophil count (ANC) ≥ 1.5/uL
* Platelets ≥ 100 x 103/uL
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present.
* Bilirubin ≤ 1.5 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dL;

  * Performance status Eastern Cooperative Oncology Group (ECOG) 0-1 or Karnofsky > 70%;
  * Men and women, ages > 18 years of age;
  * Life expectancy > 3 months;
  * Patients may have brain metastases if these are stable for at least 4 weeks and patients are not steroid dependent;
  * Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study.
* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL ]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (hCG)) within 72 hours prior to the start of study medication.Men should use avoid impregnating women during study and for 7 mos after the study.

Exclusion Criteria:

* Patients having no lesions outside the field of radiation thus nullifying the ability to measure an abscopal effect;
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic auto immune disease (e.g., rheumatoid arthritis, progressive systemic sclerosis [scleroderma]), systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis];
* Patients with a history of symptomatic interstitial lung disease OR a history of (non-infectious) pneumonitis that required oral or IV steroids or current pneumonitis.
* Patients with active HIV infection Patients with Hepatitis B and Hepatitis C infection.
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea;
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids; Tyrosine Kinase inhibitors such as erlotinib;
* Prior therapy with ipilimumab or another anti-CTLA-4 antagonist;
* Women and men who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 5mos (women) or 7mos(men) weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine New York Prebyterian hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immunotherapy + Radiation
Started | 15
Completed | 0
Not Completed | 15
Not completed — Death | 9
Not completed — Progression of disease | 6

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 65.31 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Enhance Overall Response Rate (ORR) to the Combination of Ipi/Nivo in Chemo-refractory NSCLC and Double the ORR of Ipi/RT, From 18% Based on Intent to Treat to 36%.
Description: To enhance the ORR to the combination of Ipi/Nivo in chemo-refractory NSCLC by preceding it with a combination of Ipi/RT to convert the irradiated tumor into an in situ vaccine and to double the ORR of Ipi/RT, from 18% based on intent to treat to 36%.
Time Frame: 2.5 Months, 6 Months, 3 years
Population: Participants were not assessed at 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 15
Participants
  2.5 Months | 10
  6 Months | 9
  3 Years: number analyzed (Participants) | 0

2. Secondary Outcome: Changes in T-cell Receptor (TCR) Repertoire in Peripheral Blood Are Associated With Response to Treatment
Description: changes in T-cell receptor (TCR) repertoire in peripheral blood are associated with response to treatment
Time Frame: 4 years
Population: None of the 15 enrolled subjects were enrolled at the 4 year time point.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Serum Markers IFN-b, CXCL11, sMICA, sMICB Levels/Changes Associated With Patients' Response to the Treatment.
Description: serum markers interferon-beta(IFN-B), C-X-C motif chemokine 11(CXCL11), soluble major histocompatibility complex class I-related chain A(sMICA), soluble major histocompatibility complex class I-related chain B (sMICB) levels/changes associated with patients' response to the treatment
Time Frame: 4 years
Population: None of the 15 enrolled subjects were enrolled at the 4 year time point.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

4. Secondary Outcome: Associations of Overall Response Rate (ORR) With Changes in the Microbiome
Description: associations of ORR with changes in the microbiome
Time Frame: 4 years
Population: None of the 15 enrolled subjects were enrolled at the 4 year time point.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival
Description: Patients will be followed for progression free survival.
Time Frame: 4 years
Population: None of the 15 enrolled subjects were enrolled at the 4 year time point.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Patients' Time to Progression Will be Assessed in This Study.
Description: Patients' time to progression will be assessed in this study.
Time Frame: 3 years
Population: Participants were not assessed at 3 years.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

7. Secondary Outcome: Patients' Duration of Response (DOR) Will be Assessed in This Study.
Description: Patients' duration of response (DOR) will be assessed in this study.
Time Frame: 3 years
Population: Participants were not assessed at 3 years.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival (OS)
Description: Patients will be followed for overall survival.
Time Frame: 4 years
Population: None of the 15 enrolled subjects were enrolled at the 4 year time point.
Arm/Group | Immunotherapy + Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at 2.5 months, 6 months and All-Cause mortality was assessed up to 3 years.
Description: Adverse events are documented based on the CTCAE version 5.0.
Arm/Group | Immunotherapy + Radiation
All-Cause Mortality (participants affected / at risk) | 9/15
Serious Adverse Events (participants affected / at risk) | 10/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy + Radiation (N=15)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 10 (10) — Shortness of breath
Immune mediated Hepatitis (Hepatobiliary disorders) | 1 (1) — Immune mediated Hepatitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immunotherapy + Radiation (N=15)
Abdominal distension (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 15
Abdominal Pain (Gastrointestinal disorders) | 1
acute pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 7
Alanine aminotransferase increased (Hepatobiliary disorders) | 6
Absolute Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 5
Anorexia (Gastrointestinal disorders) | 5
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Hepatobiliary disorders) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Bloating (Gastrointestinal disorders) | 2
Blood Bilirubin Increased (Hepatobiliary disorders) | 2
Blurred Vision (Eye disorders) | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Creatinine Increased (Renal and urinary disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Dysuria (Renal and urinary disorders) | 1
Edema Limbs (Vascular disorders) | 3
Eosinophilia (Blood and lymphatic system disorders) | 2
Gait disturbance (General disorders) | 1
Headache (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hoarseness (Gastrointestinal disorders) | 4
Hot Flashes (Endocrine disorders) | 2
Hyperkalemia (Blood and lymphatic system disorders) | 1
Hypercalcemia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Blood and lymphatic system disorders) | 7
Hypertension (Cardiac disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hypoalbuminea (Blood and lymphatic system disorders) | 9
Hypophysitis (Endocrine disorders) | 1
Insomnia (Nervous system disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Pain (General disorders) | 6
Peripheral Neuropathy (Nervous system disorders) | 1
Proteinuria (Investigations) | 2
Presyncope (Nervous system disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 3
Sinus Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tracheal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 1
Vertigo (Nervous system disorders) | 1
Weight Loss (Investigations) | 7

LIMITATIONS AND CAVEATS:
The study was terminated early leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT03168464/Prot_SAP_000.pdf